CLINICAL TRIAL: NCT01444729
Title: A Non-Interventional Post Approval Commitment Study To Evaluate The Outcomes Of The Various Treatment Options For Dupuytren's Contracture
Brief Title: Post Approval Commitment Study
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: B1531005
Record Dates: First submitted 2011-09-08; First posted 2011-10-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dupuytren's Contracture
Keywords: 'Dupuytren's contracture'; 'xiapex'; 'surgery'
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- xiapex: Subject treated with Xiapex
  Interventions: Drug: Xiapex
- Surgery: Fasciotomy or fasciectomy
  Interventions: Procedure: surgery

INTERVENTIONS:
Drug: Xiapex — Xiapex administration will follow SMPC
  Groups: xiapex
Procedure: surgery — Non-pharmacological treatment
  Groups: Surgery

SUMMARY:
An agreement has been made to conduct a post-approval commitment study that provides supplementary information relating to the use of Xiapex® as well as other non-pharmacological treatments for Dupuytren's contracture by health care professionals in a real world clinical setting.

DETAILED DESCRIPTION:
phase 4, open label, multi-center, prospective non-interventional descriptive

ELIGIBILITY:
Inclusion Criteria:

* Adults with a palpable cord eligible for the treatment of Dupuytren's contracture

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adults with a palpable cord eligible for the treatment of Dupuytren's contracture
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
clinical treatment success as assessed by goniometry | an expected average of 5 weeks
treatment satisfaction using the Patient or Physician Global Assessment and Satisfaction questionnaires | an expected average of 5 weeks

SECONDARY OUTCOMES:
Treatment option as determined by treating physician in consultation with patient | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, Study Director — Endo
Locations (7):
- Norway (2):
  - Auxilium Investigational Site, Bergen
  - Auxilium Investigational Site, Drammen
- Spain (5):
  - Auxilium Investigational Site, Málaga, Andalusia
  - Auxilium Investigational Site, Alcorcón, Madrid
  - Auxilium Investigational Site, Majadahonda, Madrid
  - Auxilium Investigational Site, Pamplona, Navarre
  - Auxilium Investigational Site, Valladolid